CLINICAL TRIAL: NCT00186199
Title: Determination of Voiding Patterns of Children With Vesicoureteral Reflux
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Dairiki Shortliffe, Professor Urology, Stanford University
Other Study IDs: 1790
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Vesicoureteral Reflux
Keywords: voiding patterns; flow rate; ultrasound
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine if the pattern of voiding differs in children with vesicoureteral reflux (VUR) compared to those who do not have VUR.

DETAILED DESCRIPTION:
We hope to determine the statistical difference between the flow rate and volume of urination in children with VUR compared to those without.

ELIGIBILITY:
Inclusion Criteria:

* Children with or without vesicoureteral reflux (history of VUR)
* Toilet trained and can void on command

Exclusion Criteria:

* Any voiding disorder, musculoskeletal neurologic disorders, other congenital or acquired genitourinary problems, growth disorders, recent UTI

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with history of vesicoureteral reflux, toilet trained, ambulatory, and able to void on command. Children scheduled to have procedural correction of vesicoureteral reflux
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Uroflow rate | 3 months
  Obtain pre and postoperative uroflow after VUR correction

SECONDARY OUTCOMES:
PVR | 3 months
  Pre and postoperative measures

CONTACTS AND LOCATIONS:
Overall Officials: Linda Shortliffe, MD, Principal Investigator — Department of Urology, Stanford University
Locations (1):
- Lucile Packard Childrens Hospital, Stanford, California, United States